CLINICAL TRIAL: NCT04179916
Title: Evaluation of the Physical Reaction in Immersive Virtual Reality
Brief Title: Evaluation of Physiological Reactions in Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Opole University of Technology (Other)
Collaborators: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Sebastian Rutkowski, Researcher, The Opole University of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OpoleUofTech
Record Dates: First submitted 2019-11-19; First posted 2019-11-27 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Virtual Reality
Keywords: virtual reality; VR; HRV; thermal imaging

STUDY DESIGN:
Intervention Model Description: For this study it was assumed to expose healthy volunteers for stimuli in the immersive virtual reality
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): Participants between 21 and 25 years, the Faculty of Physical Education and Physiotherapy of the Opole University of Technology Students
  Interventions: Diagnostic Test: stimulation in virtual reality

INTERVENTIONS:
Diagnostic Test: stimulation in virtual reality — HTC VIVE pro was used to stimulate patients in virtual reality. The glasses enable high resolution and high fluidity (90Hz) images to be displayed. The display used inside the glasses, OLED class, allows for accurate color replication. Numerous sensors placed in the glasses (such as gyroscope, accelerometer, magnetometer) supported by dedicated processors processing data from the sensors, instantly transfer the movement of the head of the rehabilitated person to virtual reality. Such a set allows to achieve full immersion in the virtual world. Various scenarios will be presented during the stimulation, such as beach, snow landscape, darkened room, rollercoaster ride.
  It was planned to submit 3 scenarios with a total stimulation time of up to 20 minutes.

SUMMARY:
The purpose of virtual medicine is to minimize direct contact and impact on human body during treatment. Taking into consideration the increasing accessibility of high quality electronic devices, their immense computing powers, and the continuously developing Internet infrastructure, the advancement in this area is only a matter of time. The project aims to analyze physiological reactions to stimuli in virtual reality in order to select appropriate stimulations for a group of pulmonary and cardiac patients.

DETAILED DESCRIPTION:
In recent years, the literature has shown the results of many studies undertaking the possibility of applying new technologies in rehabilitation as elements of optimization, including Virtual Reality (VR). VR can be based on computer programs that use a three-dimensional camera or sensors placed on the body to read the patient's movements and transfer them to the screen in a computer-created environment. For the most part, VR research has focused on analyzing the therapeutic potential of typical virtual games, which are not designed for clinical use, but for entertainment and relaxation.

Rehabilitation in virtual reality has also become one of the common challenges for physiotherapists and IT specialists, who develop improvement programs dedicated to various diseases and illnesses. Numerous publications are available in the scientific literature, describing the possibilities of using VR as a diagnostic and therapeutic tool. The possibility of diagnostic application of the technology in motion analysis has been demonstrated. The use of VR in the analysis of respiratory mechanics and training of pulmonary patients has also been noted. Most of the available studies concern the rehabilitation of neurological patients. There are many studies available, including meta-analyses, which confirm that the best results of rehabilitation can be achieved through the use of traditional neurological rehabilitation combined with rehabilitation conducted in virtual reality. Only few papers describe physiological reactions, including heart rate variability (HRV) and thermovision diagnostics during stimulation in immersive virtual reality.

The aim of the study is to evaluate the physiological reactions of the organism in healthy subjects during stimulation in immersive virtual reality.

This study is focused on:

Monitoring physiological parameters including heart rate variability (HRV) and thermal imaging (TI) change in healthy subjects during stimulation in immersive virtual reality.

The result of proposed research may be the answer to the following questions:

1. What changes in heart rate variability occur during the stimulation of various types of stimuli in virtual reality?
2. Which alterations in body temperature, especially in the distal parts of the upper limb, occur during stimulation in virtual reality?

The evaluation session will be conduced in the following scheme in static seated position:

1. Preparation of the research equipment
2. Measurement without stimulation in virtual reality: HRV, TI - 6 minute
3. Measurement in virtual reality: HRV, TI - simulation of cold environment (snow, wind) - 6 minute
4. Measurement in virtual reality: HRV, TI - simulation of warm environment (the beach, the sea) - 6 minute
5. Measurement in virtual reality: HRV, TI - simulation of terrifying environment (a dark room, ghosts) - 6 minute
6. Measurement without stimulation in virulent reality: HRV, TI - 6 minute
7. Completion of the measurements

ELIGIBILITY:
Inclusion Criteria:

1. Age: 21-25

Exclusion Criteria:

1. diagnosed internal diseases
2. diseases and injuries of the locomotor system impairing the function of transport, especially injuries of the upper limb
3. claustrophobia
4. eye disorders

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Thermal Imaging | 30 minutes
  The thermographic camera Flir 435-0006-03 will be used for measurements. The forearm and hand area will be observed. Photographs will be taken with a sequence of 30 seconds.

SECONDARY OUTCOMES:
Heart Rate Variability | 30 minutes
  Throughout the examination, heart rate will be monitored by the Polar H10 optical heart rate sensor. Polar H10 is a monitor armband that combines versatility, comfort and simplicity.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Rutkowski, PhD, Principal Investigator — The Opole University of Technology
Locations (3):
- San Camillo IRCCS, Venice, Italy
- Poland (2):
  - The Ministry of the Interior and Administration Hospital, Głuchołazy
  - Institute of Physiotherapy, Department of Physical Education and Physiotherapy, Opole University of Technology, Opole

IPD SHARING:
Plan to Share IPD: Yes
It was decided to provide free access to the analysed data. The data will be available upon request sent to PI: s.rutkowski@po.opole.pl.
Supporting Information: Study Protocol
Time Frame: 6 months